CLINICAL TRIAL: NCT00987584
Title: A Biologic Correlates Study for "A Phase 2 Single-Arm Study To Assess The Efficacy and Safety Of 48-Hour Continuous Intravenous Dosing Of ON 01910.Na Administered Once a Week for 3 Weeks of a 4-Week Cycle in Myelodysplastic Syndrome Patients With Trisomy 8 or Classified as Intermediate-2 or High Ris
Brief Title: Phase II Cont. IV of ON 01910.Na in MDS w/ Trisomy 8/Intermed-1, 2/High Risk
Status: Completed | Type: Observational
Sponsor: Peter L Greenberg (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor-Investigator, Peter L Greenberg, Professor Emeritus, Stanford University
Organization: Stanford University (Other)
Other Study IDs: IRB-15469; HEMMDS0023 (Other: OnCore)
Record Dates: First submitted 2009-09-24; First posted 2009-10-01 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — marrow and peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is under Molecular and Cellular Characterization of Myelodysplastic Syndromes (MDS) (eProtocol 15369). The purpose of this proposed study is to analyze existing samples taken from participants participating in a clinical trial evaluating the efficacy and safety of investigational agent ON 01910.Na (eProtocol 16214). This study will use existing blood and marrow samples to determine the rate and duration of objective hematologic and marrow responses, and duration of progression-free survival in ON01910.Na-treated MDS patients.

This study will use existing blood and marrow samples to determine the rate and duration of objective hematologic and marrow responses, and duration of progression-free survival in ON01910.Na-treated MDS patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPSS Intermediate or High risk MDS by bone marrow biopsy, marrow cytogenetics and blood counts, using FAB morphologic criteria
* Eastern Cooperative Oncology (ECOG) performance status of 0-2
* Adequate Liver Function, as evidenced by a serum bilirubin less or equal to 1.5 times the laboratory normal range (except for patients with a confirmed diagnosis of Gilberts Disease) or an ALT and AST 3 times the laboratory normal range
* A serum creatinine concentration less or equal to 2mg/dl
* Subjects must be equal or greater than 18 years of age at the time of obtaining informed consent
* Written informed consent

Exclusion Criteria:

* Prior history of leukemia or aplastic anemia
* Prior history of bone marrow transplantation
* Platelet count <100,000/mm^3

  *Prior malignancy (other than in situ cervical cancer, controlled prostate cancer, or basal cell cancer of the skin) unless treated with curative intent and without evidence of disease for greater or equal to 3 years before randomization
* Active or uncontrolled infections
* Unstable angina, congestive heart failure [NYHA>classII], uncontrolled hypertension [diastolic >100mmHg], uncontrolled cardiac arrhythmia, or recent (within 1 year) myocardial infarction
* Less than 4 weeks since receipt of any investigational product or device
* Pregnant or breast feeding
* Subjects of reproductive potential who are not using adequate contraceptive precautions, in the judgment of the investigator
* Previously enrolled in this study
* Will not be available for follow-up assessments
* Any disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of IPSS Intermediate or High risk MDS
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2009-06; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Hematologic responses | 4 months
  Marrow blast decrement

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Greenberg, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States